CLINICAL TRIAL: NCT04874012
Title: Effect of Taurine on Glycemic, Lipid and Inflammatory Profile in Individuals With Type 2 Diabetes: a Randomized Clinical Trial
Brief Title: Taurine Effect on Glycemic, Lipidic and Inflammatory Profile in Individuals With Type 2 Diabetes
Acronym: TAUGLIP-DM2
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 20200559
Record Dates: First submitted 2021-04-30; First posted 2021-05-05 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: taurine; inflammation; glucose metabolism disorders; glycated hemoglobin; diabetes mellitus, type 2; amino acids
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Inflammation; Glucose Metabolism Disorders | interventions — Taurine

STUDY DESIGN:
Intervention Model Description: Randomized, double-blind, placebo-controlled clinical trial
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The generation of the sequence of numbers will be done by a blinded researcher, after selecting the participant by the inclusion and exclusion criteria. The concealment of allocation will be implemented by a central randomization routine, conducted by researchers with access to the list and by the researcher responsible for requesting the code for placement of individuals in the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Placebo (Placebo Comparator): Participants into the placebo group will receive the same treatment regimen, but with packets of the same appearance and size containing only vehicle.
  Interventions: Other: Placebo Comparator
- Taurine (Active Comparator): Participants will receive 6 gy taurine divided into twice/day orally administration for 12 weeks.
  Interventions: Drug: Active comparator Taurine

INTERVENTIONS:
Drug: Active comparator Taurine — Participants will receive 3 g taurine, twice a day, as a powder for oral suspension (3 g/packet) for 12 weeks. Participants will be recommended to take the taurine immediately before the breakfast and dinner.
  Other Names: Taurine
  Arms: Taurine
Other: Placebo Comparator — Participants will receive the same treatment regimen and intake recommendation, but packets with the same appearance and size from those taurine ones will contain a vehicle
  Arms: Placebo

SUMMARY:
Type 2 diabetes mellitus (DM2) is characterized by chronic hyperglycemia, which is a risk factor for comorbidities and death. Although conventional pharmacotherapy is effective, some individuals do not reach the glycemic targets, requiring adjuvant therapies. Taurine is a semi-essential amino acid with antioxidant and osmoregulatory properties, commonly used as a nutritional supplement. Pre-clinical studies show its effectiveness in reducing blood glucose and cholesterol, but there are no well-conducted clinical studies evaluating the effect of taurine on glycated hemoglobin. Additionally, animal models showed that taurine had a protective effect from diabetic nephropathy. The hypothesize of this study is that taurine administration improves the glycemic, lipid, inflammatory, and anthropometric parameters in DM2 individuals.

DETAILED DESCRIPTION:
A randomized, double-blind, placebo-controlled clinical trial will be conducted at Hospital de Clínicas de Porto Alegre (HCPA), Brazil. A total of 94 participants with DM2 will be recruited and randomized on a 1:1 ratio to receive 3 g taurine as a powder for oral suspension, twice per day, for 12 weeks or packets containing placebo. Blood will be collected prior to the treatment and after 12 weeks for glycated hemoglobin, fasting glucose, insulinemia, total cholesterol and fractions, triglycerides, C-reactive protein, creatinine, urea, tumor necrosis factor-alpha (TNF-α), interleukin 1 and 6 (IL-1 and IL-6) measures. Urine will be collected at baseline and after 12 weeks for creatine, protein, and albumin measured. Anthropometric parameters and a 24-h dietary recall will be monthly investigated. Fourteen days before the end of the trial, participants will be connected to a continuous glucose monitoring system for glucose monitoring system for glucose variability evaluation. Participants will be contacted by phone weekly to report adverse effects.

ELIGIBILITY:
Inclusion criteria

* Female and male individuals, with clinical diagnosis of DM2 for at least 6 months;
* Age over 30 years;
* BMC equal to or above 18.5 kg/m2, without weight change in the last 3 months;
* HbA1c between 7.5% and 10.5%.

Exclusion criteria

* Use of herbal supplements, antioxidants, and multivitamins in the last 3 months;
* Pregnancy or lactation;
* Chronic renal failure with glomerular filtration rate calculated by MDRD < 30 mL/h;
* Myocardial infarction in the last than 6 months
* Current neoplasia;
* Chronic use of glucocorticoids;
* Bariatric surgery.

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Estimated)
Dates: Start 2021-06-12 (Actual); Primary Completion 2025-10 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
HbA1c | baseline and 12 weeks
  Changes from baseline glycated hemoglobin levels at 12 weeks

SECONDARY OUTCOMES:
Fasting glucose | baseline and 12 weeks
  Changes from baseline fasting glucose levels at 12 weeks
Insulin levels | baseline and12 weeks
  Changes from baseline insulin levels at 12 weeks
Total serum cholesterol (CT) and fractions | baseline and12 weeks
  Changes from baseline total serum cholesterol, high-density lipoprotein (HDL-C), and low-density lipoprotein cholesterol (LDL-C) levels at 12 weeks
Triglycerides serum levels | baseline and12 weeks
  Changes from baseline triglycerides serum levels at 12 weeks
Glucose variability | for 2 weeks (10-12th week)
  Changes in glucose levels throughout the day assessed by a continuous glucose monitoring system (CGMS)
Cytokine levels | baseline and 12 weeks
  Changes from baseline TNF-α, IL-1, IL-6 levels at 12 weeks
Protein creatine index | baseline and 12 weeks
  Changes from baseline protein creatinine index measured in urine at 12 weeks.
Albuminuria | baseline and 12 weeks
  Changes from baseline albuminuria levels at 12 weeks
Body mass index (BMI) | baseline and 4, 8, and 12 weeks
  Changes from baseline BMI calculated by weight (kg) and height (cm) at 4, 8, and 12 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Beatriz D Schaan, PhD, Principal Investigator — Hospital de Clínicas de Porto Alegre
Locations (1):
- Hospital de Clínicas, Porto Alegre, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Caletti G, Herrmann AP, Pulcinelli RR, Steffens L, Moras AM, Vianna P, Chies JAB, Moura DJ, Barros HMT, Gomez R. Taurine counteracts the neurotoxic effects of streptozotocin-induced diabetes in rats. Amino Acids. 2018 Jan;50(1):95-104. doi: 10.1007/s00726-017-2495-1. Epub 2017 Sep 21. PMID 28936709
- [Background] Caletti G, Olguins DB, Pedrollo EF, Barros HM, Gomez R. Antidepressant effect of taurine in diabetic rats. Amino Acids. 2012 Oct;43(4):1525-33. doi: 10.1007/s00726-012-1226-x. PMID 22302366
- [Background] Chauncey KB, Tenner TE Jr, Lombardini JB, Jones BG, Brooks ML, Warner RD, Davis RL, Ragain RM. The effect of taurine supplementation on patients with type 2 diabetes mellitus. Adv Exp Med Biol. 2003;526:91-6. doi: 10.1007/978-1-4615-0077-3_12. No abstract available. PMID 12908588
- [Background] Chan AW, Tetzlaff JM, Altman DG, Laupacis A, Gotzsche PC, Krleza-Jeric K, Hrobjartsson A, Mann H, Dickersin K, Berlin JA, Dore CJ, Parulekar WR, Summerskill WS, Groves T, Schulz KF, Sox HC, Rockhold FW, Rennie D, Moher D. SPIRIT 2013 statement: defining standard protocol items for clinical trials. Ann Intern Med. 2013 Feb 5;158(3):200-7. doi: 10.7326/0003-4819-158-3-201302050-00583. PMID 23295957
- [Background] Fukuda N, Yoshitama A, Sugita S, Fujita M, Murakami S. Dietary taurine reduces hepatic secretion of cholesteryl ester and enhances fatty acid oxidation in rats fed a high-cholesterol diet. J Nutr Sci Vitaminol (Tokyo). 2011;57(2):144-9. doi: 10.3177/jnsv.57.144. PMID 21697633
- [Background] Gomez R, Caletti G, Arbo BD, Hoefel AL, Schneider R Jr, Hansen AW, Pulcinelli RR, Freese L, Bandiera S, Kucharski LC, Barros HMT. Acute intraperitoneal administration of taurine decreases the glycemia and reduces food intake in type 1 diabetic rats. Biomed Pharmacother. 2018 Jul;103:1028-1034. doi: 10.1016/j.biopha.2018.04.131. Epub 2018 Apr 25. PMID 29710660
- [Background] American Diabetes Association. 6. Glycemic Targets: Standards of Medical Care in Diabetes-2021. Diabetes Care. 2021 Jan;44(Suppl 1):S73-S84. doi: 10.2337/dc21-S006. PMID 33298417
- [Background] American Diabetes Association. 5. Facilitating Behavior Change and Well-being to Improve Health Outcomes: Standards of Medical Care in Diabetes-2021. Diabetes Care. 2021 Jan;44(Suppl 1):S53-S72. doi: 10.2337/dc21-S005. PMID 33298416